School of Nursing

LKS Faculty of Medicine

The University of Hong Kong

Title:

New wine in old bottle: the effects of SUDOKU Mind Activation and Revitalizing Training (SMART) Program on cognitive function among people with mild cognitive impairment

document date: 2020.10.30

# THE UNIVERSITY OF HONG KONG LI KA SHING FACULTY OF MEDICINE SCHOOL OF NURSING

### **Information sheet (English version)**

## **Study Title**

New wine in old bottle: the effects of SUDOKU Mind Activation and Revitalizing Training (SMART) Program on cognitive function among people with mild cognitive impairment

# Purpose of the study

The aim of this study is to implement a SUDOKU Mind Activation and Revitalization Training (SMART) Program to promote i) cognitive health among patients with MCI, and ii) the use of active mind strategy in preventing dementia among the older adults.

#### **Target population**

For the SUDOKU Training Programme, the target population would be people with MCI as defined by a score of 19-26 out of the 30 on the Montreal Cognitive Assessment. As for the community empowerment-educational campaign, the target population will be the general public aged 55 or above.

### **Procedure**

You are invited to complete the consent form provided by research assistant to certify that they are agreed to participate in the program. A 45-minute baseline assessment including your cognitive functions, level of quality of life will then be assessed throughout face-to-face format by the research assistant. You will be randomly assigned to either Group 1 or Group 2 after the assessment.

For participants who are joining Group 1, a 24-week training including a 12-week face-to-face training session and a 12-week facilitated self-practice. The instructor will encourage and facilitate their accomplishment by giving them guidance on the taught method through regular phone call 6 times in total during self-practice period.

For participants who are joining Group 2, they are invited to join the same 24-week training after Group 1's training is completed.

Research assistant will invite the participants from Group 1 and 2 to complete the reassessment 12 and 24 weeks after the baseline assessment to capture participants' cognitive functions and level of quality of life. Research assistant will also assess the level of satisfaction to the program from Group 1 participants.

Finally, focus group interviews will be conducted to evaluate participants' satisfaction and acceptability of the program. A purposive sample of 30 participants will be interviewed in groups of six. The interview will take around 45 to 60 minutes and will be audio-taped to facilitate data analysis.

#### **Risk and Benefits**

The study intervention will not cause any pain, discomfort or harm to you.

#### Fees for participation and remuneration

You will not be charged and receive any remuneration in this program.

# Anonymity, confidentially and nature of participation

All the collected data will be subject to strict anonymity and confidentiality. Your name will not appear on any data record sheets. They will be locked up in a secure location and only the researcher can have access. All the data will also be destroyed after use. Your participation is voluntary. You may refuse to participate or may withdraw consent and discontinue the participation in the study at any time. Your decision will not affect the quality of present or future care you receive in the hospital.

#### Inquiry

This study is undertaken by Prof. Doris YU. For any inquiry, please feel free to contact Prof. YU at 39176319.

Should you have any enquiries about the rights of participant of this research study, please contact the Institutional Review Board of The University of Hong Kong/ Hospital Authority Hong Kong West Cluster at 22554086

You are cordially invited to participate in this study.

# THE UNIVERSITY OF HONG KONG LI KA SHING FACULTY OF MEDICINE SCHOOL OF NURSING

### **Informed consent form**

### Study Title:

New wine in old bottle: the effects of SUDOKU Mind Activation and Revitalizing Training (SMART) Program on cognitive function among people with mild cognitive impairment

I hereby agree to participate in the above studies. I understand that the information obtained in the study will be used for future research and maybe published in academic literature.

I also know that if I disagree with the information obtained in the public study, I can continue to participate in the study. However, all personal data is kept strictly confidential and will not be made public. I understand all the benefits and risks associated with this study.

The researcher has explained the study to me in detail and asked me to ask questions and get a satisfactory reply. If I am involved in this study and cause any physical discomfort or emotional fluctuations, the researcher will treat or refer to my treatment. I will not waive any legal rights by signing this consent form.

I hereby sign this consent form to prove that all the information provided by me is correct.

I understand that participation in this study is voluntary and I may withdraw this consent at any time without any reason, without affecting my current and future treatment.

I understand that my identity will be treated confidentially. I also allow the Institutional Review Board of the University of Hong Kong / Hospital Authority Hong Kong West Cluster and the relevant statutory bodies to directly check my research data to verify the relevant clinical research data, subject to the appropriate regulations and legislation and without infringing my privacy. (Contact number: 22554086)

| Ву | my signature below, I certify that: |
|---|---|
| | I agreed to participate this research |
| | I agreed to participate in the focus group interview and audio taped under the |
| principle of strict anonymity | |

| Name of Participant | Signature | Date |
|----------------------------|-----------|----------|
| Name of Witness | Signature | Date |
| Name of Research Assistant | Signature | <br>Date |